CLINICAL TRIAL: NCT00054015
Title: A Phase II Study of 3-Aminopyridine-2-Carboxaldehyde Thiosemicarbazone (3-AP, Triapine) in Patients With Advanced Prostate Cancer
Brief Title: 3-AP in Treating Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269675; VION-CLI-024; MCC-13110; MCC-IRB-100798
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2004-04

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

INTERVENTIONS:
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of 3-AP in treating patients who have advanced prostate cancer that has been previously treated with hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with advanced hormone-refractory prostate cancer treated with 3-AP.
* Determine the toxic effects of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive 3-AP IV over 2 hours on days 1-4. Treatment repeats every 2 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2-3 months for up to 1 year.

PROJECTED ACCRUAL: Approximately 13-27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hormone-refractory metastatic prostate cancer by one of the following methods:

  * Measurable disease
  * PSA level of at least 5 ng/mL with a positive bone scan
* Objective evidence of progressive metastatic disease in the past 3 months defined by any of the following:

  * An increase in PSA value of at least 25% (minimum absolute increase of 5 ng/mL) on at least 2 successive occasions, at least 2 weeks apart
  * A new symptomatic lesion on bone scan
  * A new metastases not in bone
  * Growth of existing non-bone measurable metastatic disease NOTE: An increase in pain or symptoms alone without other evidence of progression, or elevation of PSA or serum alkaline phosphatase alone without evidence of metastatic disease is not sufficient
* Prior bilateral orchiectomy or other primary hormonal treatment with evidence of treatment failure

  * Patients with no prior bilateral orchiectomy must have a testosterone level less than 50 ng/mL and must continue leuteinizing hormone-releasing hormone therapy while on study
* No known active CNS metastases (excluding prior CNS metastases with currently stable disease after treatment )

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL (transfusion allowed)

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* ALT/AST no greater than 5 times upper limit of normal
* Albumin greater than 2.5 g/dL
* Chronic hepatitis allowed

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No myocardial infarction within the past 3 months
* No unstable angina
* No uncontrolled arrhythmias
* No uncontrolled congestive heart failure

Pulmonary

* No dyspnea at rest

Other

* Nutrition adequate (caloric intake considered adequate for maintenance of weight)
* Fertile patients must use effective contraception
* No prior or concurrent malignancies except for non-metastatic basal cell or squamous cell skin cancer or any stage I malignancy curatively resected more than 5 years ago
* No active uncontrolled infectious process
* No other life-threatening illness
* No peripheral neuropathy greater than grade 2

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 2 weeks since prior biologic therapy

Chemotherapy

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No more than 1 prior chemotherapy regimen for metastatic disease

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since other prior hormonal therapy including any of the following:

  * Megestrol
  * Finasteride
  * Herbal products known to decrease PSA levels (e.g., saw palmetto and PC-SPES)
  * Systemic corticosteroids
* At least 4 weeks since prior flutamide therapy (6 weeks for bicalutamide or nilutamide) with continued evidence of progressive disease documented by at least 1 PSA value after discontinuation

Radiotherapy

* At least 8 weeks since prior radiopharmaceuticals (strontium chloride Sr 89, samarium Sm 153 lexidronam pentasodium)
* At least 4 weeks since prior radiotherapy and recovered

Surgery

* See Disease Characteristics
* At least 3 weeks since prior major surgery and recovered

Other

* No other concurrent investigational agents
* No other concurrent anticancer treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-12; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Sznol, MD, Study Chair — Vion Pharmaceuticals
Locations (2):
- United States (2):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida